## Title: The Outcome of Sports Vision Training on Collegiate Softball Players

NCT number: Not assigned.

Protocol ID: 2022-1225-EXP

Date: 04 Aug 2023

## SUBJECT CONSENT TO TAKE PART IN A STUDY

Investigating The Outcome of Sports Vision Training on Collegiate Softball Players and developing best practice methods for future research and sports vision training protocols.

## University of the Incarnate Word

Dear Prospective Participant: I am Kim Woideck and I am part of the UIW Sports and Vision Enhancement Service conducting this study entitled "The Outcome of Sports Vision Training on Collegiate Softball Players." You are being asked to take part in this study because you are a member of the UIW Softball Team and have been recommended by your coaches to complete sports vision training.

Female subjects: Pregnant women or nursing mothers are allowed to participate in this study. If you have personal history of epilepsy or seizures, you are not allowed to participate.

Purpose of the study: This study is designed to gather information regarding the effect of sports vision training, with goals to improve visual performance and skills. The results from this study may lead to establishing best practice methods for sports vision protocols and developing future studies.

Experimental procedures: You will be asked to participate in weekly 30-45 -minute sports vision training sessions which will include training activities designed to increase eye-hand coordination, peripheral vision awareness, reaction time, visualization, concentration, depth perception, anticipation, and low contrast perception. These training activities will be conducted by optometrists or trained optometry students under the supervision of an optometrist. For example, we will be using the Dynavision light board. This light board has 64 light buttons spanning from central to peripheral areas of the board, all within arm's reach. At random, one light will appear red. After you press the light, another random light will turn red. Your task is to press as many of the red lights as you can during the span of one minute. Another activity will include the use of Senaptec strobe glasses. These are designed to block and unblock your vision at controlled and regular intervals. These will be used during tossing, catching drills to enhance anticipation, concentration, and visualization. We will take baseline measurements through an evaluation at the Sports and Vision Enhancement Service clinic. Tests that measure visual acuity, or your ability to discern objects/letters, will be performed as well as testing your depth perception, focus flexibility, and reaction time among others. A questionnaire will then be used to investigate your overall visual performance in your sport. This questionnaire covers areas relating to visual concentration, depth perception, focusing

ability, and eye-hand coordination among other. It consists of 25 questions that you will answer and or rate on a double-sided sheet of paper.

Discomfort and risk: No additional risk is expected during your participation in this study, however some activities have the potential to produce temporary eye strain at the beginning of sports vision training. Symptoms of eye strain could include, eyes feeling tired or achy, watery, blurry vision, and/or sensitivity to light. Symptoms should be temporary, i.e. resolving in less than 2 hours. If you experience eye strain and have any questions or concerns, please address it with the doctors in vision training. Your decision to take part in the study is voluntary. You are free to choose not to take part in the study or to stop taking part at any time. If you choose not to take part or to stop at any time, it will not affect your future vision exams at Rosenberg School of Optometry. Your participation and results will not affect your status as a student athlete at UIW. First aid services are available, and all investigators are trained in CPR.

Benefits and compensation: No compensation will be provided.

Confidentiality: Everything we learn from you in the study will be confidential and your personal information and data will not be identifiable. Your evaluation and training results will be kept in a secured file cabinet. Your identity will be encrypted and efforts will be made to minimize any risks related to invasion of privacy and breach of confidentiality. If we publish the results of the study, you will not be identified in any way. It may be possible with a small cohort conducted during a specific time frame (2022) at one university that publicly accessed UIW sport information could be used to conclude which athletes may have been participants in this study. You should understand that records of your participation in the study may only be disclosed according to law, including the Federal Privacy Act, 5 U.S.C. 552a and its implementing regulations.

Entitlements: You should understand that entitlements to medical care and/or compensation in the event of injury are governed by laws and regulations, and that if you desire further information contact the Dean of the Rosenberg School of Optometry (210-883-1196). If an unanticipated event, such as a vision disorder or ill health, precludes your participation in the study, you will be informed. If you are not competent at the time to understand the nature of the event, such information will be brought to the attention of your next of kin.

Participation: The decision to participate in this study is completely voluntary. No one shall have coerced or intimidated you into participating in this activity. You should be participating because of your desire to assist the UIW Rosenberg School of Optometry in advancing the frontiers of scientific knowledge and understanding. The principal investigator and/or associate

investigator has (have) adequately answered any and all questions you may have about the study, your participation, and the procedures involved. Understand that the principal investigator and/or associate investigator will be available to answer any questions concerning procedures throughout this study. Understand that if significant new findings develop during the course of this research, which may relate to your decision to continue participation, you will be informed. Furthermore, understand that you may withdraw this consent at any time, and discontinue further participation in the study, without any prejudice to your entitlements or standing in the Rosenberg School of Optometry and University. If you decide to participate, please sign and return this consent form. If you have questions now, feel free to ask us. If you have additional questions later or you wish to report a problem that may be related to this study, you may contact me or my co-investigators, Dr Allan McCleary at amcclear@uiwtx.edu, Dr Allison Cronin at achinn@uiwtx.edu, Dr Amy Ferguson at aferguso@uiwtx.edu, Dr Chris Putnam at cputnam@uixtx.edu or Dr Lyndsey Ferris at Iferris@uiwtx.edu. The University of the Incarnate Word committee that reviews research on human subjects, the Institutional Review Board, will answer any questions about your rights as a research subject (210-829-2759—Dean of Graduate Studies and Research). You will be given a copy of this letter to keep. Thank you in advance for your cooperation and support. Sincerely, Kim Woideck, Rosenberg School of Optometry, UIW 9725 Datapoint Dr. San Antonio, TX 78229 Phone: 1 (304) 668-1026/e-mail: woideck@uiwtx.edu.

Your signature indicates that you (1) consent to take part in this research study, (2) that you have read and understand the information given above, and (3) that the information above was explained to you.

| Volunteer printed name and age |
|---------------------------------------------|
| Volunteer signature and date |
| Volunteer email |
| Investigator (informant) printed name |
| Investigator (informant) signature and date |
| Witness printed name |
| Witness signature and date |